CLINICAL TRIAL: NCT03042377
Title: The Clinical Comparative Evaluation Of Postoperative Pain In Single-Visit And Multiple-Visit Pretreatment Cases: A Prospective Randomized Clinical Trial
Brief Title: Postoperative Pain in Single-visit and Multiple-visit Retreatment Cases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Keziban Olcay, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Pain; Root Canal Infection; Endodontic Disease
Keywords: Endodontics; Retreatment; Postoperative Pain; Visual Analogue Pain Scale
MeSH Terms: conditions — Pain, Postoperative; Dental Pulp Diseases | interventions — Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: The patients were assigned to four medication groups randomly with an equal allocation rate between groups.The patients in the groups had same characteristics.
Who Masked: Participant
Masking Description: The patients were unaware as to which study group they had been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single-Visit Retreatment (Active Comparator): Root canal retreatment were performed according to the guidelines for single-visit endodontic treatments.
  Interventions: Other: Single-Visit Retreatment
- Multiple-Visit-"Calcium Hydroxide" (Active Comparator): Root canal retreatment were performed according to the guidelines for multiple-visit endodontic treatments.
  Interventions: Drug: Multiple-Visit-"Calcium Hydroxide"
- Multiple-Visit-"Corticosteroid Paste" (Active Comparator): Root canal retreatment were performed according to the guidelines for multiple-visit endodontic treatments.
  Interventions: Drug: Multiple-Visit-"Corticosteroid Paste"
- Multiple-Visit-"Antibiotic Paste" (Active Comparator): Root canal retreatment were performed according to the guidelines for multiple-visit endodontic treatments.
  Interventions: Drug: Multiple-Visit-"Antibiotic Paste"

INTERVENTIONS:
Other: Single-Visit Retreatment — The teeth in this group were treated according to the guidelines for root canal retreatment in single-session. The filling was removed and cavity was opened. Then root canal filling was removed from the root canals completely using retreatment kit. After irrigation protocol, root canals were obturated with gutta percha and coronal restoration was made using composite and/or fully crown if necessary.
  Other Names: Single-Visit Root Canal Therapy
  Arms: Single-Visit Retreatment
Drug: Multiple-Visit-"Calcium Hydroxide" — The teeth in this group were treated according to the guidelines for root canal retreatment in multiple-session. The filling was removed and cavity was opened. Then root canal filling was removed from the root canals completely using retreatment kit. After irrigation protocol, root canals were treated with calcium hydroxide and the cavity was filled with temporary restorative material.
  Other Names: Calcium Hydroxide
  Arms: Multiple-Visit-"Calcium Hydroxide"
Drug: Multiple-Visit-"Corticosteroid Paste" — The teeth in this group were treated according to the guidelines for root canal retreatment in multiple-session. The filling was removed and cavity was opened. Then root canal filling was removed from the root canals completely using retreatment kit. After irrigation protocol, root canals were treated with corticosteroid & antibiotic paste and the cavity was filled with temporary restorative material.
  Other Names: Ledermix Paste
  Arms: Multiple-Visit-"Corticosteroid Paste"
Drug: Multiple-Visit-"Antibiotic Paste" — The teeth in this group were treated according to the guidelines for root canal retreatment in multiple-session. The filling was removed and cavity was opened. Then root canal filling was removed from the root canals completely using retreatment kit. After irrigation protocol, root canals were treated with an antibiotic paste and the cavity was filled with temporary restorative material.
  Other Names: Triple Antibiotic Paste
  Arms: Multiple-Visit-"Antibiotic Paste"

SUMMARY:
The purpose of this randomized clinical trial was to evaluate the incidence of postoperative pain after retreatment using different techniques. Patients whom need retreatment were included. The presence of postoperative pain was assessed after retreatment cases at 1, 6, 12, 24 and 48 hrs.

DETAILED DESCRIPTION:
The aim of this clinical study was to evaluate the intensity and duration of postoperative pain after single-visit and multiple-visit root canal retreatment procedures. Patients who have asymptomatic failed endodontically treated teeth were included in this study and routine channel treatment procedure will be applied to these teeth. All of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. Eighty asymptomatic teeth were randomly participated into four treatment groups in terms of intracanal medicament applied. The presence of postoperative pain was assessed after 1, 6, 12, 24 and 48 hrs. Postoperative pain was recorded by each patient by using visual analogue pain scale. Before the retreatments, the nature of the study, complications and associated risks were totally explained and written informed consent was obtained from all study participants. The patients were offered local anesthetic before the treatment start. The routine root canal retreatment procedure was applied. Different intracanal medicaments used between sessions in accordance to the manufacturers' instructions. At the end of retreatment, each patient was given an evaluation sheet, explained the treatment procedure and using of visual analogue pain scales, and informed to be returned during the following one week. After one week the teeth was examined according to for pain intensity, percussion & palpation sensitivity, swelling, analgesic intake and clinical status.

ELIGIBILITY:
Inclusion Criteria:

Patients who were not included the study who;

* were pregnant or breast feeding during the duration of the study,
* have systemic disease,
* have any pain and/or any facial swelling, abscess,
* were immunocompromised,
* were under 18 yrs. and over 65 yrs. age,
* were taking antibiotics or corticosteroids within previous three months,
* have multiple teeth that required retreatment at the same time period; for eliminating pain referral,
* have root canals that could not be well-treated with orthograde retreatment.

Exclusion Criteria:

The patients who forgot to fill out the form and took antibiotics and/or analgesics right after the first appointment of the therapy were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain after Retreatment at 48 hours. | Baseline, 1, 6, 12, 24 and 48 hours.
  The primary outcome measure of the study was to assess if different intracanal medicaments and single-visit root retreatment influence the occurrence of postoperative pain.Postoperative pain was assessed using a well defined Heft-Parker visual analogue scale (VAS) scale. Each patient recorded the pain level on a 170-mm VAS scale experimental basis for revising the graphic rating scale for pain in well-defined categories at 5 time intervals as 1, 6, 12, 24 and 48 hours after treatment.The mm marks were removed from the scale and the scale was divided into 4 categories: No pain or faint pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 54 mm. Mild pain included the descriptors of weak and mild pain. Moderate pain was defined as greater than 54 mm and less than 144 mm. Intense pain was defined as equal to or greater than 144 mm. Intense pain included the descriptors of strong, severe, and maximum possible.

CONTACTS AND LOCATIONS:
Overall Officials: Keziban Olcay, DDS. PhD., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No